CLINICAL TRIAL: NCT04062786
Title: Postoperative Renal Failure in Cardiac Surgery PMSF-PVC Gradient Study
Acronym: PMSF-PVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7294
Record Dates: First submitted 2019-07-11; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Scheduled Heart Surgery; Valve Replacement; Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pmsf-PVC gradient measurement — implementation of standard standard hemodynamic monitorin

SUMMARY:
Acute renal failure is a frequent and severe postoperative complication of cardiac surgery performed under extracorporeal circulation.

It is an independent risk factor for mortality and significantly increases the length of hospital stay.

The origin of renal insufficiency after extracorporeal circulation is multifactorial (long duration of extracorporeal circulation, hemodynamic instability per and post-extracorporeal circulation, prolonged hypotension, transfusion ...).

Nevertheless, an entirely different pathophysiological mechanism, though not recent, is less often mentioned but shows renewed interest. This is the concept of renal venous congestion which may be responsible for impaired renal function in the absence of cardiac dysfunction. Based on Guyton's circulatory model, the investigators approach this systemic venous hypertension through the measurement of the Pmsf-PVC gradient.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* subject having signed an informed consent
* scheduled heart surgery:

  * Valve replacement
  * Coronary artery bypass

Exclusion Criteria:

* Any urgent surgery or redux
* Severe preoperative chronic renal failure (stage III) defined by GFR <30ml / min
* Existence of rhythm disorders (permanent ACFA) or serious cardiac conduction disorders, patients with Pacemaker
* Preoperative alteration of left ventricular ejection fraction with LVEF <40%
* Major haemodynamic instability with refractory shock defined by dobutamine ≥10μg / kg / min and / or norepinephrine ≥ 1μg / kg / min and / or epinephrine ≥ 0.2μg / kg / min.
* Intra-aortic versus assisted pelvic balloon
* Contraindication to femoral arterial catheterization
* Subject under the protection of justice, subject under guardianship or under tutorship
* Impossibility of giving the subject informed information (subject in emergency situation, difficulties in understanding the subject)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major patient with scheduled heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Evolution of the gradient Pmsf (arm) -PVC | 24 hours
  Monitor the evolution of the Pmsf (arm) -PVC gradient at H24 and compare this gradient between the two patient populations (with and without postoperative acute renal failure)

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided